CLINICAL TRIAL: NCT05993156
Title: Effects of Modified Fixed Twin Block Versus Removable Twin Block on Skeletal Class 2 Growing Patients With Mandibular Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar yousry mahmoud mostafa, primary investigator, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-3-23
Record Dates: First submitted 2023-07-06; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Malocclusion; Angle Class II; Mandible Small
Keywords: orthodontics; orthopedics; myofunctional appliance; Twinblock
MeSH Terms: conditions — Malocclusion; Malocclusion, Angle Class II; Micrognathism

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial Parallel group, two arm, equivalent trial with 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Removable twin block group (Active Comparator): participants would receive conventional removable twin block for correction of class II malocclusion for 9 months
  Interventions: Device: removable twin block
- Fixed twin block group (Experimental): participants would receive a modified fixed twin block for correction of class II malocclusion for 9 months
  Interventions: Device: modified Fixed twinblock

INTERVENTIONS:
Device: modified Fixed twinblock — modified fixed twin block functional appliance, with cemented bands on the first molars
  Other Names: F.T.B.
  Arms: Fixed twin block group
Device: removable twin block — Conventional Removable Clark twin block myofunctional appliance
  Other Names: R.T.B.
  Arms: Removable twin block group

SUMMARY:
Effects of modified fixed twin block versus removable twin block on skeletal class 2 growing patients with mandibular deficiency:

A Randomized Clinical Trial

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the effects of the modified fixed TB on class 2 growing cases and to compare its effect to the conventional removable TB

Research question Does the modified fixed twin block have the same effects as removable twin block during treatment of skeletal class 2 growing patients with mandibular deficiency?

PICO P: Growing skeletal class 2 patients with deficient mandible I : Modified Fixed Twin block C: Conventional removable Twin block

O :

Primary outcome:

Overjet

Secondary outcome:

Soft tissue Profile Antro-posterior mandibular position Mandibular length Antro-posterior maxillary position Upper and lower Incisors inclinations Durability of the appliance Patient Acceptance

Hypothesis:

There is no difference between the modified fixed or removable Twin block appliance regarding overjet reduction, dentoskeletal effects and patient perception.

8. Trial design: Randomized Clinical Trial Parallel group, two arm, equivalent trial with 1:1 allocation ratio.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal Class 2 malocclusion cases (ANB ≥ 5 degrees)
* Overjet ≥ 5 mm
* Growing patients (CVMS 3 or 4)

Exclusion Criteria:

* Skeletally mature patients 15 years old or above
* Patients with normal mandible and only protruded upper incisors.
* Syndromic, cleft patients and patients with dental anomalies
* Previous orthopaedic or orthodontic treatment
* No sex predilection.

Ages: 9 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Over jet reduction | 9 months
  the horizontal distance between upper and lower incisors

SECONDARY OUTCOMES:
Effective mandibular length | 9 months
  distance from condylon to the Pogonion points
lower incisor inclination | 9 months
  inclination of lower incisors on the mandibular plane

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
results and statistical data would be published and IPD would be available upon request

REFERENCES:
- [Background] Alhammadi MS, Halboub E, Fayed MS, Labib A, El-Saaidi C. Global distribution of malocclusion traits: A systematic review. Dental Press J Orthod. 2018 Nov-Dec;23(6):40.e1-40.e10. doi: 10.1590/2177-6709.23.6.40.e1-10.onl. PMID 30672991
- [Background] Burhan AS, Nawaya FR. Dentoskeletal effects of the Bite-Jumping Appliance and the Twin-Block Appliance in the treatment of skeletal Class II malocclusion: a randomized controlled trial. Eur J Orthod. 2015 Jun;37(3):330-7. doi: 10.1093/ejo/cju052. Epub 2014 Oct 8. PMID 25296729
- [Background] Caldwell S, Cook P. Predicting the outcome of twin block functional appliance treatment: a prospective study. Eur J Orthod. 1999 Oct;21(5):533-9. doi: 10.1093/ejo/21.5.533. PMID 10565094
- [Background] Clark William J., Mahony Derek, 2018. heal talk A journal of clinical dentistry 11.
- [Background] Clark WJ. The twin block technique. A functional orthopedic appliance system. Am J Orthod Dentofacial Orthop. 1988 Jan;93(1):1-18. doi: 10.1016/0889-5406(88)90188-6. No abstract available. PMID 3422118
- [Background] Cozza P, Baccetti T, Franchi L, De Toffol L, McNamara JA Jr. Mandibular changes produced by functional appliances in Class II malocclusion: a systematic review. Am J Orthod Dentofacial Orthop. 2006 May;129(5):599.e1-12; discussion e1-6. doi: 10.1016/j.ajodo.2005.11.010. PMID 16679196
- [Background] Ehsani S, Nebbe B, Normando D, Lagravere MO, Flores-Mir C. Short-term treatment effects produced by the Twin-block appliance: a systematic review and meta-analysis. Eur J Orthod. 2015 Apr;37(2):170-6. doi: 10.1093/ejo/cju030. Epub 2014 Jul 22. PMID 25052373
- [Background] Elfeky HY, Fayed MS, Alhammadi MS, Soliman SAZ, El Boghdadi DM. Three-dimensional skeletal, dentoalveolar and temporomandibular joint changes produced by Twin Block functional appliance. J Orofac Orthop. 2018 Jul;79(4):245-258. doi: 10.1007/s00056-018-0137-1. Epub 2018 Apr 16. PMID 29663034
- [Background] Linjawi AI, Abbassy MA. Dentoskeletal effects of the forsus fatigue resistance device in the treatment of class II malocclusion: A systematic review and meta-analysis. J Orthod Sci. 2018 Feb 15;7:5. doi: 10.4103/jos.JOS_80_17. eCollection 2018. PMID 29765917
- [Background] Matthaios S, Tsolakis AI, Haidich AB, Galanis I, Tsolakis IA. Dental and Skeletal Effects of Herbst Appliance, Forsus Fatigue Resistance Device, and Class II Elastics-A Systematic Review and Meta-Analysis. J Clin Med. 2022 Nov 26;11(23):6995. doi: 10.3390/jcm11236995. PMID 36498570
- [Background] O'Brien K, Wright J, Conboy F, Sanjie Y, Mandall N, Chadwick S, Connolly I, Cook P, Birnie D, Hammond M, Harradine N, Lewis D, McDade C, Mitchell L, Murray A, O'Neill J, Read M, Robinson S, Roberts-Harry D, Sandler J, Shaw I. Effectiveness of early orthodontic treatment with the Twin-block appliance: a multicenter, randomized, controlled trial. Part 1: Dental and skeletal effects. Am J Orthod Dentofacial Orthop. 2003 Sep;124(3):234-43; quiz 339. doi: 10.1016/S0889540603003524. PMID 12970656
- [Background] Thiruvenkatachari B, Harrison JE, Worthington HV, O'Brien KD. Orthodontic treatment for prominent upper front teeth (Class II malocclusion) in children. Cochrane Database Syst Rev. 2013 Nov 13;(11):CD003452. doi: 10.1002/14651858.CD003452.pub3. PMID 24226169